CLINICAL TRIAL: NCT05177237
Title: A Single-arm Phase II Study of Endostar Combined With Corticosteroid for Treatment of Radiation-induced Brain Necrosis in Nasopharyngeal Carcinoma
Brief Title: Endostar Combined With Corticosteroid for Treatment of Radiation-induced Brain Necrosis in Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-RN-001
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Endostar; Radiation-induced Brain Necrosis; Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endostar combined with Methylprednisolone (Experimental): Endostar combined with Methylprednisolone lasts for 10 weeks
  Interventions: Drug: Endostar

INTERVENTIONS:
Drug: Endostar — Endostar: 210 mg (14 PCS) continuous infusion for 168h, Q3W, 4 cycles. Methylprednisolone: 80mg intravenously, once daily, for 3-5 days, gradually reduced to 10mg/ day oral maintenance dose.
  Other Names: Re-human endostain

SUMMARY:
To evaluate the effectiveness and safety of Endostar combined with corticosteroids on Radiation-induced Brain Necrosis in Nasopharyngeal Carcinoma patients.

detailed description:

DETAILED DESCRIPTION:
This was a single-arm, open-label study. We aimed to evaluate the effectiveness and safety of Endostar combined with corticosteroids on Radiation-induced Brain Necrosis in Nasopharyngeal Carcinoma patients. Magnetic resonance imaging (MRI) was performed pre- and post-treatment to define the radiographic response.The primary outcome was a 2-month response rate as determined by MRI and clinical symptoms. All of the patients were followed up with for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically proven Nasopharyngeal Carcinoma(WHO 2003 I-III) .
* Presence of at least one measurable target lesion (RECIST rules) in a non irradiated region;
* age ≥18 years;
* radiation therapy history for histologically confirmed NPC administered≥6 months prior to study entry;
* radiographic evidence to support the diagnosis of RN with out tumor recurrence or metastases;
* patients had never received Antiangiogenic agents for RN treatment prior to the screening;
* patients had never received corticosteroids for RN treatment prior to the screening;
* no evidence of very high intracranial pressure suggestive of a brain hernia requiring surgery routine laboratory studies including urinalysis, complete blood count, liver function, renal function, and coagulation test within a normal range;
* to understand and be willing to sign a written informed consent.

Exclusion Criteria:

* Other types of Nasopharyngeal Carcinoma;
* Recurrent nasopharyngeal carcinoma, resection of encephalopathy, metastasis, hepatitis, other malignant tumors, neurovascular diseases, or other diseases of the nervous system;
* Inadequately controlled diabetes (FBG > 10mmol/L) and hypertension(systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg);
* Other severe concurrent disorders that occurred before enrollment (severe or unstable angor, NYHA class 3 or 4 congestive heart failure, Myocardial infarction occurred within 6 months before enrollment；Aortic dissection aortic aneurysm.) active central nervous system hemorrhage;
* pregnant or lactating women, women who have not undergone a pregnancy test (within 14 days prior to initial administration), and pregnant women;
* Patients with a history of severe mental illness or communication disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
ORR | All of the patients were followed up with for 6 months.
  2-month response rate as determined by MRI and clinical symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaochang Gong, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Yes